CLINICAL TRIAL: NCT02978898
Title: CD180 Overexpression in Follicular Lymphoma Is Restricted to the Lymph Node Compartment
Brief Title: CD180 Overexpression in Follicular Lymphoma
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0564
Record Dates: First submitted 2016-08-29; First posted 2016-12-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-08

CONDITIONS: Follicular Lymphoma
Keywords: Follicular Lymphoma; flow cytometry; CD180; Toll-like receptor; lymphoproliferative disease
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Using a multiparameter FCM approach, biologists have assessed CD180 mean fluorescence intensity (MFI) in lymph nodes (LNs) and peripheral blood (PB) samples obtained from patients with follicular lymphoma (FL; LN/PB, n544/n515), chronic lymphocytic leukemia (CLL, n526/n521), mantle cell lymphoma (MCL, n513/n517), and marginal zone lymphoma (MZL, n516/n512). Specimens from non-tumoral PB and LN (n58/n512) were used as controls.

GROUPS / COHORTS (2):
- LN Lymph nodes: Samples obtained from patients with :
  LF: Follicular lymphoma MCL: Mantle cell lymphoma CLL/SLL: chronic lymphocytic leukemia/small lymphocytic leukemia MZL : splenic marginal zone Clt :control B-cells
- PB peripheral blood: Samples obtained from patients with :
  LF: Follicular lymphoma MCL: Mantle cell lymphoma CLL/SLL: chronic lymphocytic leukemia/small lymphocytic leukemia MZL : splenic marginal zone Clt :control B-cells

SUMMARY:
Background:Altered Toll-like receptor (TLR) expression levels and/or mutations in its signaling pathway (such as MyD88 mutation) contribute to the pathogenesis of lymphoproliferative disorders (LPD). CD180 is an orphan member of the TLR family that modulates the signaling of several TLRs, but only limited studies have evaluated its expression by flow cytometry (FCM) in LPD.

Methods: Using a multiparameter FCM approach, biologists have assessed CD180 mean fluorescence intensity (MFI) in lymph nodes (LNs) and peripheral blood (PB) samples obtained from patients with follicular lymphoma (FL; LN/PB, n=44/n=15), chronic lymphocytic leukemia (CLL, n=26/n=21), mantle cell lymphoma (MCL, n=13/n=17), and marginal zone lymphoma (MZL, n=16/n=12). Specimens from non-tumoral PB and LN (n=8/n=12) were used as controls.

ELIGIBILITY:
Inclusion Criteria:

* Samples from patients with:

  * LF: Follicular lymphoma
  * MCL: Mantle cell lymphoma
  * CLL/SLL: chronic lymphocytic leukemia/small lymphocytic leukemia
  * MZL : splenic marginal zone
  * Clt :control B-cells

Exclusion Criteria:

* Patient <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 99 LN (lymph nodes) and 65 PB (peripheral blood) samples obtained from patients diagnosed with LPDs in our institution between 2012 and 2014 were evaluated for CD180 expression by FCM. The diagnosis were made according to the WHO 2008 classification, including clinical and morphological analysis, immunophenotyping, and conventional and molecular cytogenetics (and/or fluorescent in situ hybridization). The diagnoses were follicular lymphoma (FL) (LN, n=44; PB, n=15), small lymphocytic lymphoma/chronic lymphocytic leukemia (SLL)/CLL (LN, n=26; PB, n=21), MCL (LN, n=13; PB,n=17), and MZL (LN, n=16; PB, n=12). All PB samples presented circulating neoplastic B-cells, and in several cases, the diagnosis was made at the same time in LN and PB FL, n=4; SLL/CLL, n=18; MCL, n=5. MZL, n=6.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Immunophenotype Analysis by Flow Cytometry of lymph nodes samples at inclusion | At inclusion, day 0.
  Using a multiparameter FCM approach, biologists assessed the CD180 expression by our routine antigen panel in LN suspensions as well as in PB samples. Samples were analyzed on a BD FACSCanto II cytometer (BD FACS DIVA software; Becton Dickinson, San Jose, CA).
Immunophenotype Analysis by Flow Cytometry of peripheral blood samples at inclusion | At inclusion, day 0.
  Using a multiparameter FCM approach, biologists assessed the CD180 expression by our routine antigen panel in LN suspensions as well as in PB samples. Samples were analyzed on a BD FACSCanto II cytometer (BD FACS DIVA software; Becton Dickinson, San Jose, CA).

REFERENCES:
- [Result] Mestrallet F, Sujobert P, Sarkozy C, Traverse-Glehen A, Callet-Bauchu E, Magaud JP, Salles G, Baseggio L. CD180 overexpression in follicular lymphoma is restricted to the lymph node compartment. Cytometry B Clin Cytom. 2016 Sep;90(5):433-9. doi: 10.1002/cyto.b.21331. Epub 2015 Dec 11. PMID 26482097